CLINICAL TRIAL: NCT02604056
Title: Ontario Appropriate Prescribing Demonstration Project: Pragmatic, Cluster-Randomized Clinical Trial to Reduce Antipsychotic Medication Prescribing in Long-Term Care Homes
Brief Title: Pragmatic Cluster Trial for Nursing Home Antipsychotic Prescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Ontario Medical Association (Other); Health Quality Ontario (Other); Centre for Effective Practice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MOHLTCAPDP
Record Dates: First submitted 2015-11-05; First posted 2015-11-13 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Adverse Effect of Other Antipsychotics and Neuroleptics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Audit + Feedback (Active Comparator): 'Usual care' / standard quality improvement supports (including online Audit and Feedback reports for each prescriber in the home)
  Interventions: Behavioral: Audit + Feedback
- Audit + Feedback + Educational Outreach (Experimental): 'Active/full' intervention (featuring Educational Outreach offered to each prescriber and team members in the home)
  Interventions: Behavioral: Audit + Feedback; Behavioral: Audit + Feedback + Educational Outreach

INTERVENTIONS:
Behavioral: Audit + Feedback — Online Audit + Feedback practice reports detailing prescribing performance for this class of medication for each prescriber in the nursing home. (Details: http://www.hqontario.ca/Quality-Improvement/Practice-Reports/Primary-Care)
Behavioral: Audit + Feedback + Educational Outreach — The Educational Outreach program will be delivered by academic detailers, health professionals (often nurses or pharmacists) who have received specific intensive training to support prescribing providers in a particular environment, in this case long-term care homes, to make the best or appropriate clinical decisions as possible. It is defined as: "an innovative method of service-oriented educational outreach for front-line clinicians. It combines the interactive, one-on-one communication approach of industry detailers with the evidence-based, non-commercial information of academia." The Educational Outreach will be delivered in addition to online Audit + Feedback practice reports, which detail prescribing performance for this class of medication for each prescriber in the nursing home.
  Arms: Audit + Feedback + Educational Outreach

SUMMARY:
Two arm, pragmatic, cluster-randomized trial, with nursing homes allocated to the full, active intervention (featuring educational outreach offered to each prescriber and team members in the home) or standard quality improvement supports (including online audit and feedback reports for each prescriber in the home). The 'standard' quality improvement supports represent 'usual care' as these are to be launched province-wide; a concurrent control arm with no exposure to a quality improvement intervention is not feasible.

DETAILED DESCRIPTION:
The Ministry of Health and Long-Term Care and Ontario Medical Association have initiated a project aiming to improve appropriateness of prescribing in long-term care facilities (aka nursing homes) through integrated educational supports for nursing home prescribers, inter-professional care teams, as well as residents and family members. The first focus of the project is appropriate prescribing of antipsychotic medications. Working with Health Quality Ontario, the policy makers have determined that all prescribers will have the opportunity to review practice reports detailing their prescribing performance for this class of medication (aka audit and feedback).

The primary question of this pragmatic, cluster-randomized trial is: What is the effect of adding educational outreach compared to the 'usual' quality improvement supports (i.e. audit and feedback) on prescribing of antipsychotic medications in long-term care?

Secondary questions include the following:

i. What is the effect of the intervention on acute care utilization (e.g., emergency room) rates? ii. What is the effect of the intervention on incidence of patient clinical outcomes and/or adverse effects associated with antipsychotic medications (e.g., falls, aggressive behaviours)? iii. What is the effect of the interventions on medications that might be used as alternatives to antipsychotic medications (e.g., benzodiazepines)? iv. What is the cost-benefit, focusing on prescribing outcomes?

Process evaluation questions include the following:

1. How and why do the interventions work as observed?
2. Was the intervention implemented as desired in nursing homes?
3. What were the contextual factors associated with implementation?
4. Do the interventions affect precursors of behaviour (e.g., motivation, capability)?

ELIGIBILITY:
Inclusion criteria:

* Nursing homes within pre-determined regions of Ontario that expressed an interest in the full intervention (the regions, or hubs, contain a wide variety of nursing home types within a reasonable travel distance [i.e., <100 km])
* Nursing homes within the hubs in which the medical and administrative leads agree to and support the project

Exclusion criteria:

* Nursing homes with a previous or ongoing involvement in externally supported quality improvement initiatives focusing on antipsychotic medications
* Nursing homes without any prescribers caring for at least 10 residents routinely
* Nursing homes with fewer than 30 residents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Antipsychotic dispensing | 6 months post-intervention
  Number of days with antipsychotic prescriptions in the last week (count, range 0 - 7)

SECONDARY OUTCOMES:
Antipsychotic prescribing | 3 and 6 months post-intervention
  Any antipsychotic prescription during the past month (dichotomous)
Mean Antipsychotic dose | 3 and 6 months post-intervention
  Dose equivalent of antipsychotic dispensed in the past month (continuous)
Benzodiazepine (or sedative) prescribing | 3 and 6 months post-intervention
  Any prescription during the past month (dichotomous)
Anti-depressant prescribing | 3 and 6 months post-intervention
  Any prescription during the past month (dichotomous)
Acetaminophen prescribing | 3 and 6 months post-intervention
  Any prescription during the past month (dichotomous)
Difficulty in performing activities | 3 and 6 months post-intervention
  Activities of Daily Living long form scale (continuous variable, range 0-28)
Aggressive behaviour scale | 3 and 6 months post-intervention
  Extent of aggressive behaviour (continuous variable, range 0-12)
Pain | 3 and 6 months post-intervention
  Pain scale (continuous variable, range 0-3)
Depression | 3 and 6 months post-intervention
  Depression rating scale (continuous variable, range 0-14)
Falls | 3 and 6 months post-intervention
  Number of falls in the past month (count)
Emergency Room visits | 3 months post-intervention
  Number of ER visits during the previous 3 months (count)
Hospitalizations | 3 months post-intervention
  Number of hospital visits visit during the previous 3 months (count)

CONTACTS AND LOCATIONS:
Overall Officials: Noah Ivers, Principal Investigator — Family Doctor and Research Scientist

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tadrous M, Fung K, Desveaux L, Gomes T, Taljaard M, Grimshaw JM, Bell CM, Ivers NM. Effect of Academic Detailing on Promoting Appropriate Prescribing of Antipsychotic Medication in Nursing Homes: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2020 May 1;3(5):e205724. doi: 10.1001/jamanetworkopen.2020.5724. PMID 32453383
- [Derived] Desveaux L, Saragosa M, Rogers J, Bevan L, Loshak H, Moser A, Feldman S, Regier L, Jeffs L, Ivers NM. Improving the appropriateness of antipsychotic prescribing in nursing homes: a mixed-methods process evaluation of an academic detailing intervention. Implement Sci. 2017 May 26;12(1):71. doi: 10.1186/s13012-017-0602-z. PMID 28549480
- [Derived] Desveaux L, Gomes T, Tadrous M, Jeffs L, Taljaard M, Rogers J, Bell CM, Ivers NM. Appropriate prescribing in nursing homes demonstration project (APDP) study protocol: pragmatic, cluster-randomized trial and mixed methods process evaluation of an Ontario policy-maker initiative to improve appropriate prescribing of antipsychotics. Implement Sci. 2016 Mar 29;11:45. doi: 10.1186/s13012-016-0410-x. PMID 27026584